CLINICAL TRIAL: NCT05880784
Title: Peer Coaching and Clinical Audit to Facilitate Implementation of the Package of Essential Non-Communicable Diseases (PEN) in Nepal: a Mixed Method Implementation Study
Brief Title: PEN Implementation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shahid Gangalal National Heart Centre (Other)
Collaborators: Kathmandu University School of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: PEN Study
Record Dates: First submitted 2023-04-28; First posted 2023-05-30 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Package of Essential Non-Communicable Diseases (PEN); Peer Coaching; Clinical Audit; Mixed Method Implementation Study
MeSH Terms: interventions — Clinical Audit; Methods

STUDY DESIGN:
Intervention Model Description: The study is being conducted in public (primary level) health facilities with at least one PEN-trained staff in the Bhaktapur district in Nepal. The seventeen health facilities were randomized into control and intervention groups. Randomization was conducted in excel using the RAND function. Out of 17, nine facilities were categorized into intervention groups and the remaining eight into control groups. The intervention consists of peer coaching and clinical auditing processes reinforcement to promote a team-based care approach for NCD management in the health facilities.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Practice (Placebo Comparator): Eight primary healthcare centers in the Bhaktapur district of Nepal will be selected as a control group. The centers will be assessed for the baseline PEN service evaluation and at the end of one year, evaluation will be performed again in the centers for any change in the PEN services.
  Interventions: Other: Continuation of usual practice without intervention
- Peer coaching and clinical audit (Active Comparator): Nine primary healthcare centers in the Bhaktapur district of Nepal will be selected as an intervention group. The centers will be assessed for the baseline PEN service evaluation and then will be provided the peer coaching and clinical audit sensitization within 6 months of the intervention period. At the end of one year, an evaluation will be performed again in the centers for any change in the PEN services.
  Interventions: Other: Reinforcement of Peer coaching and clinical audit

INTERVENTIONS:
Other: Reinforcement of Peer coaching and clinical audit — The goal of the proposed research study is to test the effectiveness and feasibility of an intervention to enhance peer coaching and clinic audit activities to facilitate the implementation of the Package of Essential Non- Communicable Diseases (PEN) in Nepal.
  Arms: Peer coaching and clinical audit
Other: Continuation of usual practice without intervention — No intervention will be carried out, instead usual practice will be evaluated at the start and the end of the study period.
  Arms: Usual Practice

SUMMARY:
There is a gap in the implementation of PEN services as well as in the monitoring and evaluation of the WHO PEN in Nepal. One reason for such gaps is due to a lack of team-based care in low-resource settings like Nepal. Both peer coaching and clinical audit have been shown to be cost-effective ways to improve NCD care. However, no data is available regarding its implementation and outcome. Besides, there is a lack of a proven module of peer coaching and clinical audit for effective NCD care implementation. To address this gap, the investigators designed an intervention to reinforce peer coaching and clinical audit practices in health facilities to improve WHO PEN implementation for better NCD management in Nepal.

Aims of Implementation Research

* To assess implementation outcomes (acceptability, adoption, feasibility, penetration, cost and sustainability) of onsite-peer coaching and clinical audit reinforcement intervention on PEN Program implementation at primary healthcare centers.
* To evaluate the effectiveness of onsite-peer coaching and clinic audit reinforcement intervention in PEN program delivery at health facilities.
* To identify barriers and enabling factors impacting the adoption of onsite-peer coaching and clinical audit in the implementation of the PEN program.

DETAILED DESCRIPTION:
Non-communicable diseases (NCDs) kill approximately 41 million people each year. Over 80% of all premature deaths include NCD-related deaths, such as deaths from cardiovascular diseases (17·9 million deaths annually), cancers (9·3 million), respiratory diseases (4.1 million), and diabetes (2.0 million). Eighty percent of these deaths occur in low- and middle-income countries (LMIC). In Nepal, 51% of all deaths were due to NCDs in 2018. Effective prevention and management to curb mortalities and morbidities from NCDs are possible - and, are widely being implemented. Early detection and management remain central to NCD control.

For early detection and management of NCDs and to prevent life-threatening complications, a cost-effective intervention through an integrated approach, the World Health Organization (WHO) Package of Essential Noncommunicable Diseases Interventions (WHO PEN) was developed. The package provides a holistic guide, including guidelines on screening, diagnosis, treatment and referral processes of NCD patients for early detection and management of chronic diseases within the community with a systematic approach to strengthen the primary health care system.

Furthermore, NCD care is impacted by significant gaps in the capacity of health institutions and systems in terms of training, and availability of adequate resources, including human resources and supplies of necessary medicines. To cope with the shortages of healthcare workers in LMICs, primary care systems can include team-based care strategies according to the WHO PEN strategy.

One of the key aspects of the PEN package to promote NCD management is team-based care. Due to the shortage of physicians and health workers in most countries in the South East and South Asian region, team-based care strategies are added as an integral component of the WHO PEN package. Team-based care is advised in order to provide effective and continuous patient-centered care. WHO PEN package team-based care includes peer coaching and clinical audit.

WHO PEN was introduced in Nepal in 2016 with the main aim to increase access to NCD-related services in the primary health centers and health posts under the Multi-Sectoral Action Plan for NCD Prevention and Control (2014-2020). Nepal Government developed its own PEN Protocol based on WHO PEN Package to promote NCD management. It consists of four protocols for the prevention of heart attack, strokes and kidney disease through integrated management of diabetes and hypertension; health education and counseling on healthy behaviors; prevention of Chronic Obstructive Pulmonary Disease (COPD) and Asthma; and screening and referral of suspected breast and cervical cancer at Primary Health Center (PHC) level. PEN was initially piloted in two districts and expanded to additional 16 districts in 2018. At present primary Cardiovascular Disease (CVD) care using WHO PEN is only available in health facilities in 30 (out of a total of 77) districts.

ELIGIBILITY:
Inclusion Criteria:

* public (primary level) health facilities with at least one PEN-trained staff in Bhaktapur district in Nepal.

Exclusion Criteria:

* public (primary level) health facilities without at least one PEN-trained staff in Bhaktapur district in Nepal.
* public (primary level) health facilities in other districts in Nepal.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Acceptability of Intervention Measure 4-item questionnaire | 6 months
  Higher score indicate higher acceptability. Score will range from 1 to 5 with Scores 4 and 5 representing higher scores and scores 1 and 2 will represent lower scores. Higher scores will represent better acceptability.
Acceptability of the intervention by peer coaches and other health facility staff | 6 months
  Codes and themes from Qualitative Interviews to capture insights, experiences and satisfaction of health facility staff
Completion of peer coaching activities/ orientation | 6 months
  Number of staff who completed peer coaching orientation/ training. Data abstraction from Pre-post evaluation of checklist for supportive supervision & monitoring
Clinical audits performed | 6 months
  Number of clinical audits performed (or, Number of clinical audit form filled). Data abstraction from clinical audit documents
Completeness of clinical audit form | 12 months
  Clinical audit scores at 3, 6 and 12 months. Data abstraction from clinical audit documents
Proportion of health facility staff involved in implementation of PEN protocol and routine clinical audits | 6 months
  Number of health facility staff implementing PEN protocol and routine clinical audit activities/ Number of total health facility staff engaged in patient care activities.
  Routine observation and data abstraction from clinical audit document
Time taken to perform a clinical audit activities | 6 months
  Time spent to complete a single clinical audit activity. Time spent for clinical audit activities in a month
  Routine observation and data abstraction from clinical audit document
Health facility staff re-oriented and trained for PEN protocol implementation | 6 months
  Number of staff re-oriented to conduct peer coaching, plus Number of staff trained by the peer coaches and involved in PEN protocol implementation.
  Data abstraction from training and intervention evaluation document form
Additional cost-incurred for peer coaching activities | 6 months
  Cost of intervention package development and training. Additional time for clinical auditing. Data abstraction from financial report; cost estimation for the time and resource involved in health facility
Additional cost for clinical auditing | 6 months
  Cost of intervention package development and training. Additional time for clinical auditing. Data abstraction from financial report; cost estimation for the time and resource involved in health facility
Willingness to continue peer-coaching and clinical audit activities for PEN program implementation and adherence to PEN after intervention duration | 6 months
  Qualitative Interviews with peer-coaches and health facility staff

CONTACTS AND LOCATIONS:
Overall Officials: Dipanker Prajapati, MBBS, MD, Principal Investigator — Shahid Gangalal National Heart Centre, Kathmandu, Nepal
Locations (1):
- Shahid Gangalal National Heart Centre, Kathmandu, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: No
The quantitative data of the study will include the pre and post-test scores and Likert scale scoring of the Acceptability of Intervention Measure 4-item questionnaire. These data will be included in the study result section. The individual site information and the details of the qualitative and quantitative analysis will be presented in the results section itself after data analysis.